CLINICAL TRIAL: NCT03663946
Title: Drug Use Investigation on Combination Therapy With Yervoy and Opdivo (Unresectable or Metastatic Renal Cell Carcinoma)
Brief Title: A Study to Observe the Onset of Immune-related Adverse Reactions in Patients With Non-surgical or Renal Cell Carcinoma (RCC) That Has Spread
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8MK
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients taking combination therapy with Yervoy and Opdivo: Medical records will be reviewed for safety and treatments for specific ADR
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Patients with non-surgical or renal cell carcinoma that has spread who are starting treatment for the first time with Yervoy and Opdivo in the real world

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic renal cell carcinoma who are initiating treatment for the first time with Yervoy and Opdivo in accordance with the Japanese package insert will be included in this PMS

Exclusion Criteria:

* Patients receiving combination therapy with Yervoy and Opdivo for non RCC indication will be excluded from this PMS

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unresectable or metastatic renal cell carcinoma who are initiating treatment for the first time with Yervoy and Opdivo
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of immune-related AE's | Approximately 13 weeks
Incidence of immune related SAE's | Approximately 13 weeks

SECONDARY OUTCOMES:
Incidence of treatment for immune-related adverse reactions | Approximately 13 weeks
Incidence of unknown AE's | Approximately 13 weeks
Incidence of unknown SAE's | Approximately 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm